CLINICAL TRIAL: NCT01512173
Title: A Randomised, Double Blind, Controlled, Multicentre Study in Infants With Infantile Hemangioma to Compare Propranolol Gel to Placebo.
Brief Title: Study in Infants With Infantile Hemangioma to Compare Propranolol Gel to Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00400 GL 2 01 1A; 2011-003144-50 (EudraCT Number)
Record Dates: First submitted 2012-01-06; First posted 2012-01-19 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Infantile Hemangioma
Keywords: Propranolol gel; Hemangioma; capillary neoplasm; vascular tissue; neoplasm by histologic type; neoplasm; therapeutic uses; pharmacologic actions; adrenergic beta-antagonists; adrenergic antagonist; adrenergics agent; neurotransmitter agent; molecular mechanism of pharmacological action; physiological effects of drugs
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- propranolol gel (Experimental)
  Interventions: Drug: propranolol gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: propranolol gel — Topical administration twice daily
  Arms: propranolol gel
Drug: Placebo — Topical administration twice daily
  Arms: Placebo

SUMMARY:
There is an unsatisfied medical need for a first-line treatment of localized uncomplicated proliferating Infantile Hemangioma with a good benefit/risk profile.

Pierre Fabre Dermatologie has developed a new formulation of propranolol (V0400 GL 01A) which is a topical gel adapted to paediatric use.

The objective of this study is to evaluate topical propranolol efficacy and safety in the management of localized hemangioma.

ELIGIBILITY:
Main Inclusion Criteria:

* only one proliferating Infantile Hemangioma present anywhere on the body except on the head, the neck, the hands and on the diaper area, with largest diameter diameter ≥ 1cm and ≤ 5 cm.

Main Exclusion Criteria:

* more than one Infantile Hemangioma with largest diameter ≥ 1cm
* medically unstable health status that may interfere with his/her ability to complete the study
* Infantile Hemangioma requires, according to Investigator's judgment, a systemic treatment
* the patient has previously been administered treatment for IH or surgical and/or medical procedures (e.g. laser therapy) have been performed to treat the IH

Ages: 35 Days to 150 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Complete/nearly complete resolution of the Infantile Hemangioma at week 12. | week 12
  Complete/nearly complete resolution of the Infantile Hemangioma at week 12 compared to baseline

SECONDARY OUTCOMES:
On-site parent(s) or guardian(s) qualitative assessments of efficacy | week 2 , week 4, week 8, week 12 and week 24
  categorical endpoints for Infantile Hemangioma evolution (4-points scale)
Persistence of efficacy 12 weeks after the end of treatment | Week 24
  Persistence of complete/nearly complete resolution of the Infantile Hemangioma at week 24 compared to week 12.
Safety profile (descriptive analysis of AE) | Day 0, week 2, week 4, week 8, week 12 and week 24
Local tolerance of the propranolol gel(description over time by treatment group) | week 2, week 4, week 8 and week 12

CONTACTS AND LOCATIONS:
Locations (17):
- France (9):
  - CHU Bordeaux Hôpital Pellegrin-Enfants - Unité de Dermatologie pédiatrique, Bordeaux
  - Hôpital Saint Vincent de Paul - Dermatologie Pédiatrique, Lille
  - CHU Lyon Est Hôpital mère enfant - Consultation des angiomes, Lyon Bron
  - CHU Timone - Service de dermatologie, Marseille
  - Hôpital Mère-Enfant - Service de Néonatologie et Réanimation Pédiatrique, Nantes
  - CHU Necker enfants malades - Service de dermatologie, Paris
  - CHU Saint-Etienne Hôpital Nord - Service de dermatologie, Saint-Etienne
  - CHU Toulouse Hôpital des enfants - Département cardio-pédiatrique, Toulouse
  - Hôpital de Clocheville - Centre de Pédiatrie Gatien, Tours
- Poland (3):
  - Pomorskie Centrum Traumatologii im. M. Kopernika w Gdańsku Klinika Chirurgii i Urologii Dzieci i Młodzieży GUMed, Gdansk
  - Uniwersytet Medyczny w Łodzi Klinika Chirurgii i Onkologii Dziecięcej, Lodz
  - Instytut "Pomnik-Centrum Zdrowia Dziecka", Klinika Onkologii, Warsaw
- Spain (5):
  - Hospital Sant Pau de Barcelona, Barcelona
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia